CLINICAL TRIAL: NCT05930600
Title: Internal Jugular Venous Distensibility Index and Innominate Venous Flow Patterns As Predictors of Response to Fluid Administration in Elective Surgery Patients
Brief Title: Internal Jugular Venous Distensibility Index and Innominate Venous Flow Patterns As Predictors of Fluid Responsiveness
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Principal investigator, MD, PhD, Anesthesiologist Consultant, Indonesia University
Other Study IDs: IndonesiaUAnes044
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Fluid Responsiveness; Hemodynamic Monitoring
Keywords: Internal Jugular Venous Distensibility Index; Innominate Venous Flow Patterns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Ultrasonography of Internal Jugular Vein — Non invasive monitoring of fluid responsiveness
Device: Doppler Echocardiograhy — Non invasive monitoring of fluid responsiveness

SUMMARY:
The measurement of internal jugular vein distensibility index corresponds to the measurement of stroke volume using trans-thoracic Doppler echocardiography in assessing the response to fluid administration in elective surgical patients.

ELIGIBILITY:
Inclusion Criteria:

1. Utilizing intraoperative mechanical ventilation with a tidal volume of 8 ml/kg (PBW).
2. ASA physical status 1-3.
3. Mongoloid ethnicity.
4. Willing to participate in the research and sign the informed consent.

Exclusion Criteria:

1. Patients with symptoms and signs of fluid overload, such as pulmonary edema, pleural effusion, ascites, and peripheral edema.
2. Patients with chronic or acute kidney dysfunction, renal replacement therapy history, and/or oliguria (urine output <0.5 ml/kg/hour).
3. Patients with cardiovascular diseases, including heart failure, cardiac arrhythmias, moderate-to-severe valvular abnormalities, a history of angina/myocardial infarction, pulmonary hypertension, and peripheral artery disease.
4. Patients with anatomical abnormalities in the neck and chest region that make it impractical to perform jugular vein ultrasound and transthoracic echocardiography.
5. Jugular vein thrombosis.
6. Superior vena cava syndrome.
7. Placement of jugular vein catheter.
8. Body mass index (BMI) greater than 30.0 kg/m2.
9. Patients with contraindications to the use of muscle relaxants.
10. Patients with lung hyperinflation and pleural effusion.

Drop out criteria:

1. Patients who wish to withdraw from the study.
2. Post-anesthesia induction complications and emergencies.
3. Transthoracic echocardiography provides a less representative image due to difficult acoustic window.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-65 years undergoing elective surgery with general anesthesia at RSUPN dr. Cipto Mangunkusumo Jakarta.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
IJV distensibility index correlation to fluid responsiveness | 1 day
  Correlation between IJV distensibility index and fluid responsiveness defined as increase of stroke volume more than 10% after fluid challenge

SECONDARY OUTCOMES:
Comparison of IJV distensibility index in fluid responders and non-fluid responders. | 1 day
Detection of sensitivity, specificity, positive predictive value, negative predictive value, and best cut off value of IJV distensibility index to predict fluid responsiveness | 1 day
  By ROC curve and Youden index
Correlation of IJV distensibility index and stroke volume | 1 day
Innominate vein flow velocity correlation to fluid responsiveness | 1 day
  Correlation between Innominate vein flow velocity and fluid responsiveness defined as increase of stroke volume more than 10% after fluid challenge

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, Principal Investigator — Indonesia University
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia